CLINICAL TRIAL: NCT01693055
Title: Safety and Efficacy Evaluation of UltheraTM in Treatment of Baggy Eyelid,Phase 4.
Brief Title: Safety and Efficacy Evaluation of UltheraTM in Treatment of Baggy Eyelid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ulthera, Inc (Industry)
Responsible Party: Principal Investigator, Chan-Yeong Heo, Assistant professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-1207/162-004; L-2012-408-3 (Other Grant/Funding Number: JOYMG Co.,Ltd)
Record Dates: First submitted 2012-09-18; First posted 2012-09-26 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Orbital Fat Prolapse
Keywords: orbital Computed Tomography; baggy eyelids; orbital fat prolapse; UltheraTM; high intensity focused ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UltheraTM (Experimental): UltheraTM 100 shots (infraorbital region 30shots, lateral orbital region 40shots, upper eyelid 30 shots) on the Rt, and Lt periorbital area, respectively using 1.5mm and 3.0mm probe
  Interventions: Device: UltheraTM 100 shots

INTERVENTIONS:
Device: UltheraTM 100 shots — UltheraTM 100 shots (infraorbital region 30shots, lateral orbital region 40shots, upper eyelid 30 shots) on the Rt, and Lt periorbital area, respectively using 1.5mm and 3.0mm probe

SUMMARY:
Study title

* Safety and Efficacy Evaluation of UltheraTM in Treatment of Baggy Eyelid Study design
* single arm and Investigator Initiative pilot study

ELIGIBILITY:
Inclusion Criteria:

* Age >20 years, Age < 50 years
* people who want to improve baggy eyelid
* Information consent obtained

Exclusion Criteria:

* previous lower eyelid surgical history
* scar on lower eyelid after trauma
* bleeding tendency
* aesthetic addiction, drug abuse, alcohol abuse

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The distance from the inferior orbital rim to the skin | Change from Screening in distance at 12weeks after Ulthera treatment
  Difference between the distance ( from the inferior orbital rim to the skin) measured by orbital CT at Screening and 12weeks after UltheraTM treatment

SECONDARY OUTCOMES:
The distance from the most protrusive baggy eyelid to the orbital septum | Change from Screening in distance at 12weeks after UltheraTM treatment
  The distance(mm),from the most protrusive baggy eyelid to the orbital septum will be measured by a plastic surgeon with orbital CT films. Each participant will do Orbital CT scan 2 times, at screening and 12weeks after treatment
Subject Satisfaction for baggy lower eyelid | Change from Screening in satisfaction at 4 weeks and 12weeks
  5-point scale for Subject Satisfaction in baggy lower eyelid. The subject satisfaction is calculated as a score between 0 and 4( 0= very poor, 4= very good).
Improvement of baggy lower eyelid | Change from Screening in baggy lower eyelid at 12weeks after UltheraTM treatment
  Improvement of baggy lower eyelid will be assessed by Two plastic surgeons. Both assessors will evaluate Improvement of baggy lower eyelid including skin laxity and orbital fat prolapse using 5-point scale.
  0= no involvement
  1. mild
  2. moderate
  3. marked
  4. severe

CONTACTS AND LOCATIONS:
Overall Officials: Chanyeong Heo, Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National Univ. Bundang Hospital, Gumi-dong, Bundang-gu, Seongnam-si, Gyeonggi-do, South Korea